CLINICAL TRIAL: NCT05788016
Title: Developing and Testing an Opioid Taper Intervention Before Total Knee Arthroplasty: Phase 2 Intervention Development
Brief Title: Developing an Opioid Taper Intervention Before Total Joint Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Kevin Riggs, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-300009887; 1K23AR080224-01A1 (NIH)
Record Dates: First submitted 2023-03-02; First posted 2023-03-28 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Arthritis Knee; Arthritis Hip; Chronic Pain
Keywords: Opioids
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pharmacist-led opioid taper intervention (Experimental): The participant will attempt to taper their opioid dose by ~50% during the 4-6 week preoperative period. Participants will meet with a clinical pharmacist, who will provide some basic education on pain and opioids, and will propose an opioid taper schedule. The pharmacist will then follow-up with the participant by phone each week until surgery to assess progress and adjust the taper as necessary.
  Interventions: Behavioral: opioid taper

INTERVENTIONS:
Behavioral: opioid taper — The participant will attempt to taper their opioid dose by ~50% during the 4-6 week preoperative period

SUMMARY:
The goal of this clinical trial is to develop an pharmacist-led preoperative opioid taper intervention for patients undergoing total knee or hip replacement who are on chronic opioids before their surgery. The main questions it aims to answer are:

* Is the intervention feasible and acceptable to patients?
* Does the intervention result in a decrease in opioid dose during the preoperative period?

Participants will meet with a clinical pharmacist, who will provide some basic education on pain and opioids, and will propose an opioid taper schedule. The pharmacist will then follow-up with the participant by phone each week until surgery to assess progress and adjust the taper as necessary.

ELIGIBILITY:
Inclusion Criteria:

* decided to pursue primary, unilateral total knee or hip arthroplasty with planned surgery date in 4-8 weeks
* currently taking between 20 and 90 MME of oral opioids, and that dose has been stable for at least 3 months
* have a reliable telephone number for contact
* speaks English

Exclusion Criteria:

* Taking opioid medications that include:

  * Buprenorphine
  * Methadone
  * Long-acting formulations of opioid pain medications (e.g., extended-release oxycodone and extended-release morphine)
  * Transdermal formations of opioid pain medications (e.g., fentanyl patches)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability | From enrollment until approximately 2 weeks after surgery
  Mixed-methods assessment of the intervention by participants. Participants will provide qualitative feedback at multiple points during and after the intervention, and will quantitatively rate satisfaction at the end of the study. These results will be analyzed jointly to determine acceptability.

SECONDARY OUTCOMES:
Study Recruitment Rate | From enrollment until approximately 2 weeks after surgery
  In order to assess feasibility of the taper intervention, we will track the proportion of participants who are offered enrollment that ultimately enroll (will be measured separately for those offered enrollment in person and those who are mailed information about the study)
Study Retention Rate | From enrollment until approximately 2 weeks after surgery
  In order to assess feasibility of the taper intervention, we will track the proportion of enrolled participants who complete the final study visit.
Taper Efficacy | From enrollment until the time of surgery
  change in opioid dose from enrollment through surgery
Perioperative Pain | From enrollment until approximately 2 weeks after surgery
  pain scores throughout the perioperative period

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R Riggs, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Hospital-Highlands, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No